CLINICAL TRIAL: NCT02567370
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single-ascending Dose Study With a Food-Effect Cohort to Evaluate the Safety, Tolerability, and Pharmacokinetics of AMG 581 in Healthy Subjects and Subjects With Schizophrenia
Brief Title: Single-ascending Dose Study With a Food-Effect Cohort to Evaluate AMG 581
Acronym: FIH
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20130100
Record Dates: First submitted 2015-09-16; First posted 2015-10-05 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2015-10

CONDITIONS: Schizophrenia or Schizoaffective Disorder
Keywords: Schizophrenia or Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- AMG 581 (Active Comparator)
  Interventions: Drug: AMG 581

INTERVENTIONS:
Drug: AMG 581 — Active drug
  Arms: AMG 581
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to find out the time it takes to absorb, distribute, breakdown and remove the drug from the body, safety and tolerability of AMG 581 in healthy participants and subjects with schizophrenia.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetic profile of single-ascending oral doses of AMG 581 in healthy subjects and subjects diagnosed with schizophrenia or schizoaffective disorder receiving antipsychotic treatment.

This will be a placebo-controlled, single-ascending oral-dose study of AMG 581 with a food-effect cohort. Approximately 70 subjects will be enrolled. This study will enroll healthy subjects into 8 cohorts (Cohorts 1,2,3,4,5,6,8 and 9), and subjects with schizophrenia or schizoaffective disorder receiving antipsychotic medication into a single cohort (Cohort 7).

ELIGIBILITY:
Inclusion Criteria:

* Provide informed consent prior to initiation of any study-related procedure
* Male and female subjects ≥ 18 to ≤ 45 years of age at the time of screening
* Non-nicotine or non-tobacco for healthy subjects
* No history of relevant medical disorders
* BMI ≥ 18.0 and ≤ 30.0
* Non-reproductive females
* Males practicing effect birth control
* Avoid tanning/direct sunlight
* Willing to consume high-fat meal
* Schizophrenia or schizoaffective disorder
* PANSS score ≤ 4 points on a few items (i.e. conceptual disorganization, hallucinatory behavior, excitement, suspiciousness/persecution, hostility, depression, anxiety, disorientation, uncooperativeness, disturbance of volition, and poor impulse control) / total score ≤ 80 points

Exclusion Criteria:

* Females lactating/breastfeeding
* Pregnant partners of male subjects
* Tremor or gait disturbance
* History of hereditary shorten QT syndrome
* Malignancy or tumor (other than skin cancers)
* History of GI disease
* QTc ≥ 450 msec or ≤ 380 msec
* Creatinine clearance < 80 mL/min at screening

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2015-08; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Reported treatment-emergent adverse events | 15 days
  Number and percent of subjects experiencing adverse events
Changes in systolic/diastolic blood pressure | 15 days
  Summaries over time and/or changes from baseline over time in systolic and/or diastolic blood pressure
Changes in heart rate | 15 days
  Summaries over time and/or changes from baseline over time in heart rate
Changes in respiratory rate | 15 days
  Summaries over time and/or changes from baseline over time in respiratory rate
Changes in temperature | 15 days
  Summaries over time and/or changes from baseline over time in temperature
Changes in ECGs | 15 days
  Summaries over time and/or changes from baseline over time in ECGs
Scores at each study visit for Simpson Angus Scale (SAS) | 15 days
  Summaries over time and/or changes from baseline over time in Simpson Angus Scale (SAS) score
Scores at each study visit and summary by cohort for Barnes Akathisia Rating Scale (BARS) | 15 days
  Summaries over time and/or changes from baseline over time in Barnes Akathisia Rating Scale (BARS) score
Subject incidence of treatment-emergent suicidal ideation and behavior as measured by Columbia-Suicide Severity Rating Scale (C-SSRS) | 15 days
  Subject incidence of treatment-emergent suicidal ideation and behavior as measured by Columbia-Suicide Severity Rating Scale (C-SSRS) summarized by cohort

SECONDARY OUTCOMES:
Peak plasma concentration (Cmax) | 15 days
  Peak plasma concentration (Cmax)
Area under the plasma concentration versus time curve (AUC) | 15 days
  Area under the plasma concentration versus time curve (AUC)
Median of tmax | 15 days
  Median of tmax

OTHER OUTCOMES:
AMG 581 metabolites in plasma | 15 days
  Metabolites of AMG 581 in plasma
Subjective experience follow administration of AMG 581 as measured by the Bond and Lader visual analogue scale (VAS) | 15 days
  To assess the subjective experience of study subjects following administration of AMG 581 as measured by the Bond and Lader visual analogue scale (VAS)
Subjective experience follow administration of AMG 581 as measured by the Positive and Negative Syndrome Scale (PANSS) | 15 days
  To assess the subjective experience of study subjects following administration of AMG 581 as measured by the Positive and Negative Syndrome Scale (PANSS; subjects diagnosed with schizophrenia or schizoaffective disorder receiving antipsychotic treatment only)
Relationship between plasma concentration of AMG 581 and QTc interval | 15 days
  To explore the relationship between changes in QTc interval (msec) and AMG 581 plasma concentration (ng/mL)
Effect of food on plasma concentration of AMG 581 | 43 days
  To assess the effect of a high-fat meal on the plasma concentration of AMG 581 (ng/mL) comparing median of tmax between fasted and fed conditions (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- Research Site, Glendale, California, United States

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com